CLINICAL TRIAL: NCT02090829
Title: Promoting Social Perceptual Learning With Oxytocin in Autism
Brief Title: Intranasal Oxytocin and Learning in Autism
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of Minnesota (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1402M48250
Record Dates: First submitted 2014-02-28; First posted 2014-03-18 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; Oxytocin; Syntocinon
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo Comparator: Intranasal Placebo Intranasal placebo The placebo is identical to the oxytocin formulation with the exception of the active compound.
  Route of administration: Intranasal Planned exposure: Each participant will receive one dose of intranasal placebo per day for 5 days.
  One dose equals 6 spray puffs (3 puffs in each nostril).
  Interventions: Other: Placebo
- Experimental Group (Active Comparator): Intranasal oxytocin (Trade name: Syntocinon) Pharmacological class: The pharmacologic and clinical properties of Syntocinon are identical with the naturally occurring hormone oxytocin, which is released from the posterior pituitary.
  Route of administration: Intranasal Planned exposure: Each participant will receive one dose of intranasal oxytocin (24 IU) per day for 5 days.
  One dose of 24 IU equals 6 spray puffs (3 puffs in each nostril). Oxytocin will be imported from Victoria Pharmacy Zurich- Switzerland.
  Interventions: Drug: Syntocinon (synthetic oxytocin)

INTERVENTIONS:
Drug: Syntocinon (synthetic oxytocin) — Syntocinon is a nine residue cyclic peptide; the hormone is prepared synthetically to avoid possible contamination with vasopressin and other small polypeptides with biologic activity.
  Other Names: Syntocinon
  Arms: Experimental Group
Other: Placebo — Placebo Comparator: Intranasal Placebo Intranasal placebo The placebo is identical to the oxytocin formulation with the exception of the active compound.
  Route of administration: Intranasal Planned exposure: Each participant will receive one dose of intranasal placebo per day for 5 days.
  One dose equals 6 spray puffs (3 puffs in each nostril).
  Arms: Placebo Group

SUMMARY:
: The objective of this study is to determine the tolerability and therapeutic potential of oxytocin in children and adolescents with Autism Spectrum Disorders (ASD) when paired with a computer game intervention that is designed to enhance face perception skills. We designate two measures as our primary outcomes, based on prior published work with these interventions, and we propose a sample based on power analyses from these prior results. A second objective of this study is to learn about the breadth of possible positive effects that this combination therapy might have for children with ASD. To this end, we include a host of other exploratory measures that assess aspects of social motivation and attention, social perception, and social cognition. Thus, a second objective is to conduct a "signal finding" study - to gather outcome data on a range of dependent variables that theoretically should be related to oxytocin's effects on social processes, but for which there are no prior data. The signal finding aspect of this study will provide the preliminary data needed to design a more targeted follow up study.

DETAILED DESCRIPTION:
This is a double-blind placebo-controlled trial of intranasal oxytocin in 52 children and adolescents with ASD. Diagnosis will be confirmed using Diagnostic and Statistical Manual (DSM) criteria, supported by the Autism Diagnostic Interview and the Autism Diagnostic Observation Schedule. Subjects will be randomized to 24 IU intranasal oxytocin or placebo for a 5 day period with concomitant game play of the FaceStation computer games, developed at CHOP. Measures of social function and cognition will be administered before and after the game play period. Two measures of social functioning will serve as our primary endpoints; all other measures will be treated as exploratory variables, with significance testing corrected for multiple comparisons.

Recognizing faces is critical to social functioning, and can be improved for individuals with ASD by using intervention software in the form of appropriately designed computer games. The effects of this type of social intervention may be amplified with the concurrent use of oxytocin. Furthermore, these learning effects may impact social skills in general and translate to the level of the individual's everyday social behavior. Thus, the objective of this study is to determine the safety and therapeutic potential of intranasal oxytocin in children and adolescents with ASD when paired with a computer game intervention that is designed to enhance face perception skills.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 12-17 years, Mental age ≥ 7 (as measured by an IQ test such as the Differential Ability Scales II).
2. Gender: males
3. Diagnosis of an ASD
4. Consent: parent/guardian permission and child assent.
5. Ability to complete tasks: adequate vision, motor control of a keyboard and mouse, and fluency in English
6. Study participant needs to be on clinically stable, in the opinion of the study clinicians. Stability will be assessed by the clinicians based on information from and conversations with the parent, if necessary. The parent needs to commit verbally to not making any changes to his or her child's current treatments for the duration of this study.

Exclusion Criteria:

1. History of traumatic brain injury, epilepsy/seizure disorder (except febrile seizures), or other significant medical, genetic, or acquired neurological abnormality affecting brain function and motor, sensory or higher cognitive functioning.
2. Patients with one or more of the following: HIV, HBV, HCV, hemophilia (bleeding problems, recent nose and brain injuries), abnormal blood pressure (hypotension or hypertension), drug abuse, immunity disorder, or severe depression.
3. Sensory impairments (e.g., significant vision/hearing loss).
4. Gestational age below 35 weeks and/or perinatal injury.
5. Profound mental retardation (e.g., IQ < 45) or sensory-motor difficulties that would preclude valid use of diagnostic instruments
6. Lack of impairment in face recognition as determined by average or above average performance on the Benton Face Recognition Task.
7. Female participants.
8. Patients who are sensitive to Syntocinon or any components of its formulation.
9. Fever at the time of the baseline visit, defined as temperature above 37.5 degrees Celsius or 99.5 degrees Fahrenheit.
10. Judgment by the study physician/P.I. (Suma Jacob, M.D,) that the patient is not suitable for the study due to unforeseeable safety issues.

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Post-testing on the The Part/Whole Identity Test | Baseline/Follow-up post testing (max 12 days)
  4) Part/Whole Identity Test measures the extent to which the participant employed a featural or holistic face recognition strategy. In this task, a sample face is presented for 4 sec, followed by a test face composed of either two whole faces or two face parts. As expected in Part/Whole Identity, effect sizes ranged from a low 0.30 for the part mouth condition to a high of 0.81 for the whole eye condition, such that the condition measuring holistic processing in the eye region was most sensitive to group differences. This measure was also most sensitive to behavioral changes with the LFI intervention trial.
Change from Baseline to Post-testing on the Reading the Mind in the Eyes Task | Baseline to Post-testing (max. 12 days)
  Reading the Mind in the Eyes Test (child version) (Baron-Cohen, et al., 2001) is a test of emotion recognition. This test asks children to pick the best word out of four options to describe the mental state of a set of eyes. The test includes 28 photographs of eyes with both affective (e.g., upset) and cognitive (e.g., thoughtful) mental state words as choices.

SECONDARY OUTCOMES:
Change from Baseline to Post-testing on measures of social attention, reward/motivation, perception and cognition | Baseline/follow-up (after max 12 days)
  Behavioral tasks: watching social interactions eye tracking-task, happy faces eye-tracking tasks, signal detection social task, discrimination task

CONTACTS AND LOCATIONS:
Overall Officials: Suma Jacob, M.D. Ph.D, Principal Investigator — University of Minnesota Department of Psychiatry
Locations (1):
- Center for Neurobehavioral Development, Minneapolis, Minnesota, United States